CLINICAL TRIAL: NCT04942613
Title: Engaging Medically Complex Veterans in Tele-Rehabilitation Using a Biobehavioral Approach: A Pilot Study of Feasibly and Acceptability
Brief Title: Engaging Medically Complex Veterans in Tele-Rehabilitation Using a Biobehavioral Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E3730-P; 21-2773 (Other: COMIRB)
Record Dates: First submitted 2021-05-26; First posted 2021-06-28 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Multimorbidity; Physical Deconditioning
Keywords: telerehabilitation; high intensity; biobehavioral; social support; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 2 groups: Group1 will receive the intervention first for 12 weeks, and Group2 will receive the waitlist control for 12 weeks. At the end of 12 weeks, Group2 will crossover to the intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Multicomponent Telehealth Intervention (Group1) (Experimental): This group will be randomized to receive the 12-week multicomponent intervention first. They will receive individual physical therapy sessions, group physical therapy sessions, and biobehavioral interventions emphasizing program engagement and increased daily physical activity. Most interventions will be provided synchronously through videoconferencing. Each participant will receive an individualized home exercise program.
  Interventions: Behavioral: Motivational Interviewing Techniques; Other: Physical Therapy Interventions; Other: Qualitative Interview
- Education (Group2) (Other): This group will be randomized to 12-week waitlist control condition. They will receive a one-hour education session every 2 weeks (6 sessions total) on general health topics (e.g., basic nutrition, stress reduction, sleep hygiene). At the end of 12 weeks, they will transition to the 12-week multicomponent intervention
  Interventions: Other: Education; Other: Qualitative Interview
- Research Participants (Other): Participants will be asked to complete up to 2 semi-structured interviews following completion of the 12-week multicomponent intervention. The first interview will occur within 3 weeks of program completion (by week 15 for Group 1 and by week 27 for Group 2). The second interview will occur between 3 to 6 months after the first interview.
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Behavioral: Motivational Interviewing Techniques — Motivational Interviewing Techniques including but not limited to open-ended questions, reflection, affirmations, and summary will be used to build participant rapport, support behavior change (physical activity), and facilitate program engagement.
  Arms: Multicomponent Telehealth Intervention (Group1)
Other: Physical Therapy Interventions — strengthening, balance, functional activities, stretching, breathing, aerobic endurance exercise
  Arms: Multicomponent Telehealth Intervention (Group1)
Other: Education — Education on general health topics which may include the following: basic nutrition, stress reduction, sleep hygiene
  Arms: Education (Group2)
Other: Qualitative Interview — Qualitative interview to explore patient perspectives of the multicomponent telerehabilitation program (physical therapy, biobehavioral interventions, technology, and social support interventions) and how they contribute to program engagement and participation as well as changes in physical activity.

SUMMARY:
The aims of this study are to determine the feasibility and acceptability of a multicomponent telerehabilitation program for medically complex older Veterans and to preliminarily assess participant outcomes (physical activity, physical function, quality of life, loneliness) to the program.

DETAILED DESCRIPTION:
The aims of this study are to determine the feasibility and acceptability of the multicomponent telerehabilitation program and to preliminarily assess participant outcomes. The multicomponent program/intervention consists of 3 core components: 1) high-intensity rehabilitation interventions, 2) biobehavioral interventions, and 3) social support. The delivery of the program is supported by various technologies allowing for synchronous and asynchronous care and monitoring. Synchronous telerehabilitation will occur individually and in virtual groups. Feasibility and acceptability will be assessed by Veteran adherence to program components and validated surveys. Preliminary responsiveness will be assessed primarily by change in 7-day average step count and secondarily by other physical function tests and patient reported outcome measures. Study findings will have immediate clinical impact as they will guide implementation of safe and effective telerehabilitation strategies for medically complex older Veterans who lack access to standard in-person rehabilitation services.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age and older
* Multiple chronic conditions (Charlson Comorbidity Index 3)
* Impaired physical function (< or = 10 repetitions on 30 second sit to stand test)

Exclusion Criteria:

* Life expectancy < 12 months
* Acute or progressive neurological disorder (e.g. Amyotrophic Lateral Sclerosis, recent stroke)
* Moderate to severe dementia without caregiver assistance (< 18 on telephone Montreal Cognitive Assessment (MoCA Blind)
* Unstable medical condition precluding safe participation in progressive rehabilitation (e.g. unstable angina)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Stevens-Lapsley, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Started | 25 | 25
Completed 12 Week Oucomes | 24 | 25
Not Completed 12 Week Outcomes | 1 | 0
Started Multicomponent Telehealth Intervention (Group 2 Only) | 0 | 25
Completed (24 week outcomes) | 20 | 22
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (6.0) | 69.9 (7.3) | 69.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 22 | 46
  Not Hispanic or Latino | 0 | 3 | 3
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 17 | 24 | 41
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Military Branch [Count of Participants; unit: Participants]
  Army | 10 | 13 | 23
  Navy | 7 | 3 | 10
  Air Force | 7 | 5 | 12
  Marines | 1 | 4 | 5
Marital Status [Count of Participants; unit: Participants]
  Married | 14 | 17 | 31
  Widowed | 1 | 2 | 3
  Divorced or Separated | 5 | 3 | 8
  Single | 5 | 2 | 7
  Cohabitating | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  High School or Equivalent | 2 | 1 | 3
  Associates Degree or Some College | 12 | 8 | 20
  Bachelors Degree | 5 | 7 | 12
  Post-baccalaureate | 6 | 9 | 15
Employment [Count of Participants; unit: Participants]
  Retired | 20 | 20 | 40
  Working (full- or part-time) | 3 | 2 | 5
  Unemployed or other | 2 | 3 | 5
Support at Home [Count of Participants; unit: Participants]
  All the time | 11 | 15 | 26
  Some or Most of the Time | 8 | 6 | 14
  No | 6 | 4 | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (6.6) | 31.0 (5.4) | 31.0 (6.0)
Functional Comorbidity Index [Mean (Standard Deviation); unit: units on a scale] — The Functional Comorbidity index (FCI) has been designed specifically in relation to physical function. It includes 18 diagnoses, counting their presence or absence, resulting in a cumulative sum score of 0 to 18. Higher scores indicate greater comorbidity burden.
  units on a scale | 6.0 (1.7) | 5.9 (2.1) | 6.0 (1.9)
Functional Comorbidity Index Top 6 Diagnoses [Count of Participants; unit: Participants] — The Functional Comorbidity index (FCI) has been designed specifically in relation to physical function. It includes 18 diagnoses, counting their presence or absence, resulting in a cumulative sum score of 0 to 18. Higher scores indicate greater comorbidity burden. These are the 6 most common comorbidities.
  Participants
    Arthritis | 16 | 17 | 33
    Obesity (BMI > 30 kg/m2 | 15 | 16 | 31
    Visual Impairment | 15 | 14 | 29
    Depression | 18 | 11 | 29
    Degenerative Disc Disease | 16 | 12 | 28
    Anxiety (Includes PTSD) | 13 | 14 | 27
Prescription Medications (total) [Mean (Standard Deviation); unit: number of prescriptions] | 14.1 (7.9) | 11.6 (5.3) | 12.9 (6.8)
Polypharmacy (≥ 5 meds) [Count of Participants; unit: Participants] | 24 | 24 | 48
Top 3 Frequent Medications [Count of Participants; unit: Participants]
  Antidepressant | 12 | 9 | 21
  Diuretic | 6 | 10 | 16
  Beta Blocker | 7 | 8 | 15
Berkman Social Disengagement Scale (disengaged) [Count of Participants; unit: Participants] — Number of participants who scored as Disengaged.
  Participants | 10 | 10 | 20
Telephone Montreal Cognitive Assessment (cognitive impairment) [Count of Participants; unit: Participants] | 6 | 10 | 16
Patient Health Questionnaire (PHQ-9) positive for depression [Count of Participants; unit: Participants] — Number of participants who scored positive for depression.
  Participants | 7 | 7 | 14
Generalized Anxiety Disorder (GAD) positive for anxiety [Count of Participants; unit: Participants] — Number of participants who scored positive for anxiety.
  Participants | 4 | 3 | 7
Mobile Device Proficiency Questionnaire (MDPQ-16) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 16-80; higher scores indicated higher ability to perform technology tasks.
  units on a scale | 67.9 (13.6) | 69.2 (9.9) | 68.5 (11.8)
Number of Rural Participants [Count of Participants; unit: Participants] — A participant was determined to be rural if their zip code for their home address was listed on the Federal Office of Rural Health Policy Eligible Zip Codes file.
  Participants | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Adherence to the Multicomponent Telehealth Intervention
Description: Adherence will be calculated as the proportion of the number of sessions attended out of the number prescribed per protocol (32 sessions)
Time Frame: Program end- 12 weeks in Intervention group (Group1); 24 weeks in Waitlist control (Group2)
Population: All participants; data from both groups will be pooled for analysis.
Measure: Median (Inter-Quartile Range); unit: Proportion of sessions attended
Units Other Than Participants: Sessions
Groups:
- All Participants: Combination of both arms
Arm/Group | All Participants
Number analyzed (Participants) | 50
Number analyzed (Sessions) | 32
Proportion of sessions attended | 0.95 [0.81 to 1.00]

2. Secondary Outcome: Physical Activity
Description: Physical activity will be measured via accelerometry and will include average 7-day step count
Time Frame: Change from pre-program (baseline for Group 1, 12 weeks for Group 2) to post-program (12 weeks for Group 1, 24 weeks for Group 2).
Population: All participants with complete step count data will be analyzed. Since only pre-program and post-program data were collected, the data were pooled to increase statistical power.
Measure: Median (Inter-Quartile Range); unit: steps
Arm/Group | All Participants
Number analyzed (Participants) | 36
steps | -95 [-514 to 915]

3. Secondary Outcome: Feasibility of the Multicomponent Telehealth Intervention
Description: Feasibility will be measured through a validated survey: Feasibility of Intervention Measure consists of 4 items rated on a 5-point Likert scale (1) completely disagree to (5) completely agree. The average of the 4 items are reported. Higher scores indicate greater feasibility of the program.
Time Frame: Program end- 12 weeks in Intervention group (Group1); 24 weeks in Waitlist control (Group2)
Population: All participants with complete data; data from both groups will be pooled for analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 50
units on a scale | 5.0 [4.8 to 5.0]

4. Secondary Outcome: Acceptability of the Multicomponent Telehealth Intervention
Description: Acceptability will be measured through a validated survey: Acceptability of Intervention Measure consists of 4 items rated on a 5-point Likert scale (1) completely disagree to (5) completely agree. The average of the 4 items are reported. Higher scores indicate greater acceptability of the program."
Time Frame: Program end- 12 weeks in Intervention group (Group1); 24 weeks in Waitlist control (Group2)
Population: All participants with complete data; data from both groups will be pooled for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 50
score on a scale | 5.0 [4.7 to 5.0]

5. Secondary Outcome: Participant Recruitment
Description: Recruitment will be tracked as part of feasibility and to inform a future trial. Recruitment will be reported as a proportion of those enrolled out of the total number screened via phone screen.
Time Frame: Baseline
Population: Number phone screened
Measure: Count of Participants; unit: Participants
Groups:
- Recruitment: Proportion of number enrolled from number completing phone screen.
Arm/Group | Recruitment
Number analyzed (Participants) | 84
Participants | 50

6. Secondary Outcome: Satisfaction of the Multicomponent Telehealth Intervention
Description: Participation satisfaction with care provided via telerehabilitation will be assessed via the VA's approved survey: V-signals. It consists of 11 items rated on a 5-point Likert scale from (1) strongly disagree to (5) strongly agree). The average of the 11 items are reported. Higher scores indicate better satisfaction.
Time Frame: Program end- 12 weeks in Intervention group (Group1); 24 weeks in Waitlist control (Group2)
Population: All participants with complete data; data from both groups will be pooled for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 50
score on a scale | 4.9 [4.6 to 5.0]

7. Secondary Outcome: Safety Event Count
Description: The Safety Event Count is the cumulative number of study related (possibly, probably, or definitely) adverse events and severe adverse events counted from baseline to program end. Events will be categorized by type
Time Frame: Program end- 12 weeks in Intervention group (Group1); 24 weeks in Waitlist control (Group2)
Population: Number of adverse events
Measure: Number; unit: number of adverse events
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 25 | 25
number of adverse events
  Falls | 2 | 1
  ED Visit | 3 | 1
  Hospitalization | 1 | 0
  Other | 1 | 3
  Unrelated Falls | 13 | 19
  Unrelated ED Visits | 7 | 10
  Unrelated Hospitalizations | 4 | 2
  Unrelated Other | 4 | 10

8. Secondary Outcome: Exercise Stages of Change Questionnaire
Description: Four-item questionnaire used to determine an individual's stage of change (pre-contemplation, contemplation, preparation, action, or maintenance)
Time Frame: Change from Baseline to 12 weeks
Population: All Participants
Measure: Count of Participants; unit: Participants
Groups:
- Multicomponent Telehealth Intervention (Group1) Baseline; Multicomponent Telehealth Intervention (Group 1) 12 Weeks: This group will be randomized to receive the 12-week multicomponent intervention first. They will receive individual physical therapy sessions, group physical therapy sessions, and biobehavioral interventions emphasizing program engagement and increased daily physical activity. Most interventions will be provided synchronously through videoconferencing. Each participant will receive an individualized home exercise program.
  Motivational Interviewing Techniques: Motivational Interviewing Techniques including but not limited to open-ended questions, reflection, affirmations, and summary will be used to build participant rapport, support behavior change (physical activity), and facilitate program engagement.
  Physical Therapy Interventions: strengthening, balance, functional activities, stretching, breathing, aerobic endurance exercise
- Education (Group2) Baseline; Education (Group 2) 12 Weeks: This group will be randomized to 12-week waitlist control condition. They will receive a one-hour education session every 2 weeks (6 sessions total) on general health topics (e.g., basic nutrition, stress reduction, sleep hygiene). At the end of 12 weeks, they will transition to the 12-week multicomponent intervention
  Education: Education on general health topics which may include the following: basic nutrition, stress reduction, sleep hygiene
Arm/Group | Multicomponent Telehealth Intervention (Group1) Baseline | Multicomponent Telehealth Intervention (Group 1) 12 Weeks | Education (Group2) Baseline | Education (Group 2) 12 Weeks
Number analyzed (Participants) | 25 | 24 | 25 | 25
Participants
  Pre-contemplation | 0 | 0 | 1 | 1
  Contemplation | 8 | 3 | 12 | 11
  Preparation | 12 | 3 | 6 | 6
  Action | 1 | 8 | 2 | 2
  Maintenance | 4 | 10 | 4 | 5

9. Secondary Outcome: Self-efficacy for Exercise (SEE) Scale
Description: Nine item questionnaire used to measure an individual's self-efficacy for exercising under different conditions. Each item is rated on a scale of 0 (not confident) to 10 (confident). The average of the 9 items is calculated; higher scores indicate better self-efficacy. The change from baseline to 12 weeks is calculated as 12 weeks minus baseline; thus, positive change scores indicate improvement in self-efficacy.
Time Frame: Change from Baseline to 12 weeks
Population: All participants completing the 12 week testing. Group 1 had 1 withdrawal and 1 participant unable to complete all outcome measures due to new medical diagnosis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 23 | 25
score on a scale | 0.0 [-2.8 to 1.0] | 0.0 [-1.8 to 1.4]

10. Secondary Outcome: 30 Second Sit to Stand
Description: The test uses a standard height chair and requires the participant to stand up and sit down as many times as possible in 30 seconds. More completions indicate better physical function.
Time Frame: Change from Baseline to 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Number of sit to stand repetitions
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 23 | 25
Number of sit to stand repetitions | 1.0 [-1.0 to 4.0] | 1.0 [0.0 to 2.0]

11. Secondary Outcome: Arm Curl Test
Description: This is a functional performance test for upper body strength and is performed on each arm (one arm at a time). It requires the participant to perform as many arm curls (biceps curls) as possible in 30 seconds. Males use an 8lb weight and females use a 5lb weight. Scores are continuous, and higher scores indicate greater arm strength (better outcome)
Time Frame: Change from Baseline to 12 weeks
Population: All participants completing the 12 week testing. Group 1 had 1 withdrawal and 1 participant unable to complete all outcome measures due to new medical diagnosis. Group 2 had 1 participant not complete this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Number of arm curl repetitions
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 23 | 24
Number of arm curl repetitions
  Dominant | 3.0 [0.0 to 5.0] | 0.5 [-1.5 to 4.0]
  Non-dominant: number analyzed (Participants) | 22 | 24
  Non-dominant | 3.0 [0.0 to 5.5] | 1 [-0.5 to 3.5]

12. Secondary Outcome: 2-minute Step Test
Description: This is a functional performance test for aerobic endurance. It requires participants to march in place for 2 minutes (alternating legs), and the score is the number of repetitions completed on the right leg. Scores are continuous, and higher scores indicate better aerobic endurance.
Time Frame: Change from Baseline to 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: number of repetitions
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 23 | 25
number of repetitions | 15.0 [7.0 to 31.0] | 0.0 [-5.0 to 15.0]

13. Secondary Outcome: Activity Measure for Post-Acute Care (AM-PAC) Basic Mobility Outpatient Routine Short Form
Description: This questionnaire consists of 18 items rated on a 4-point Likert scale from 1 (unable) to 4 (none) to address the prompt: How much difficulty do you currently have. The total score is reported by summing each item; scores can range from 18 to 72. Higher scores indicate better mobility and less impairment/disability.
Time Frame: Change from Baseline to 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 23 | 25
units on a scale | 4.0 [-2.0 to 11.0] | 1.6 [0.0 to 7.0]

14. Secondary Outcome: 3-Item Loneliness Scale
Description: This scale has three items and a simplified set of response categories that is designed to measure overall loneliness. Score range: 3-9. Higher scores indicate higher loneliness.
Time Frame: Change from Baseline to 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 23 | 25
units on a scale | 0.0 [0.0 to 1.1] | 0.0 [-1.0 to 0.0]

15. Secondary Outcome: PROMIS-29+2 Profile v2.1 Physical Health and Mental Health Subscales Only
Description: This is a patient reported outcome measure to assess physical health (subscale) and mental health (subscale). It is a 29-item questionnaire, and most items are rated on a 5-point Likert scale. There is 1 pain intensity item rated on a 0 (no pain) to 10 (worst pain imaginable) scale. PROMIS scores were transformed to a T-score where 50 represents the population mean, and the standard deviation is 10. The method reported by Hays et al. in 2018 was used to calculate the physical health and mental health subscales. Higher scores for subscales listed indicate better physical and mental health.
Time Frame: Change from Baseline to 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Multicomponent Telehealth Intervention (Group1) | Education (Group2)
Number analyzed (Participants) | 23 | 25
score on a scale
  Physical Health | 2.1 [-0.4 to 4.3] | -0.3 [-2.2 to 3.1]
  Mental Health | 0.3 [-1.8 to 7.0] | -2.1 [-6.2 to 1.6]

16. Secondary Outcome: Participant Retention
Description: Participant retention will be tracked as part of feasibility and to inform a future trial. Retention will be reported as a proportion of the total number of participants who complete all outcome measure timepoints out of the total who complete baseline measures.
Time Frame: 12 Weeks and 24 Weeks
Population: Total number of participants. The investigators considered retention to be study retention in addition to intervention retention, which included the outcome assessments at all time points. Thus, even though participants in Group 1 did not receive any intervention from weeks 12-24, they were still considered enrolled in the study until their 24 week outcome assessment was completed, they withdrew, or were lost to follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Multicomponent Telehealth Intervention (Group 1): This group will be randomized to receive the 12-week multicomponent intervention first. They will receive individual physical therapy sessions, group physical therapy sessions, and biobehavioral interventions emphasizing program engagement and increased daily physical activity. Most interventions will be provided synchronously through videoconferencing. Each participant will receive an individualized home exercise program.
  Motivational Interviewing Techniques: Motivational Interviewing Techniques including but not limited to open-ended questions, reflection, affirmations, and summary will be used to build participant rapport, support behavior change (physical activity), and facilitate program engagement.
  Physical Therapy Interventions: strengthening, balance, functional activities, stretching, breathing, aerobic endurance exercise
- Education (Group 2): This group will be randomized to 12-week waitlist control condition. They will receive a one-hour education session every 2 weeks (6 sessions total) on general health topics (e.g., basic nutrition, stress reduction, sleep hygiene). At the end of 12 weeks, they will transition to the 12-week multicomponent intervention
  Education: Education on general health topics which may include the following: basic nutrition, stress reduction, sleep hygiene
Arm/Group | Multicomponent Telehealth Intervention (Group 1) | Education (Group 2)
Number analyzed (Participants) | 25 | 25
Participants
  12 Week Retention | 24 | 25
  24 Week Retention | 20 | 22

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Multicomponent Telehealth Intervention (Group1) During and Related to Intervention; Multicomponent Telehealth Intervention (Group 1) Not During and Not Related to Intervention: This group will be randomized to receive the 12-week multicomponent intervention first. They will receive individual physical therapy sessions, group physical therapy sessions, and biobehavioral interventions emphasizing program engagement and increased daily physical activity. Most interventions will be provided synchronously through videoconferencing. Each participant will receive an individualized home exercise program.
  Motivational Interviewing Techniques: Motivational Interviewing Techniques including but not limited to open-ended questions, reflection, affirmations, and summary will be used to build participant rapport, support behavior change (physical activity), and facilitate program engagement.
  Physical Therapy Interventions: strengthening, balance, functional activities, stretching, breathing, aerobic endurance exercise
- Education (Group 2) During and Related to Multicomponent Telehealth Intervention; Education (Group 2) Not During and Not Related to Intervention: This group will be randomized to 12-week waitlist control condition. They will receive a one-hour education session every 2 weeks (6 sessions total) on general health topics (e.g., basic nutrition, stress reduction, sleep hygiene). At the end of 12 weeks, they will transition to the 12-week multicomponent intervention
  Education: Education on general health topics which may include the following: basic nutrition, stress reduction, sleep hygiene
Arm/Group | Multicomponent Telehealth Intervention (Group1) During and Related to Intervention | Education (Group 2) During and Related to Multicomponent Telehealth Intervention | Multicomponent Telehealth Intervention (Group 1) Not During and Not Related to Intervention | Education (Group 2) Not During and Not Related to Intervention
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/25 | 4/25 | 12/25 | 16/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multicomponent Telehealth Intervention (Group1) During and Related to Intervention (N=25) | Education (Group 2) During and Related to Multicomponent Telehealth Intervention (N=25) | Multicomponent Telehealth Intervention (Group 1) Not During and Not Related to Intervention (N=25) | Education (Group 2) Not During and Not Related to Intervention (N=25)
Cardiac (Cardiac disorders) | 3 (3) | 3 (3) | 2 (3) | 6 (10)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Fall (General disorders) | 2 (2) | 1 (1) | 10 (12) | 10 (19)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT04942613/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT04942613/ICF_002.pdf